CLINICAL TRIAL: NCT04976361
Title: Macular Vessels Density Before and After Panretinal Photocoagulation in Patients With Proliferative Diabetic Retinopathy
Brief Title: Macular Vessels Density Before and After PRP in Patients With Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Principal Investigator, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VD befor and after PRP
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: PRP
Keywords: OCTA; PRP

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic Patients with PDR (Experimental): PRP for each diabetic patient included in this study.
  Interventions: Other: PRP was done using visulas green laser machine (Carl Zeiss Meditec AG Geoschwitzer Str. 51-52,07745 jena, Germany)

INTERVENTIONS:
Other: PRP was done using visulas green laser machine (Carl Zeiss Meditec AG Geoschwitzer Str. 51-52,07745 jena, Germany) — PRP was done using visulas green laser machine (Carl Zeiss Meditec AG Geoschwitzer Str. 51-52,07745 jena, Germany)

SUMMARY:
In this study, OCTA is used to study the vascular changes following PRP in patients with PDR; regarding vessels density at 1 month and 6 months follow up period and measure superficial, deep, and outer retina for fovea, para-fovea and whole image.

DETAILED DESCRIPTION:
The global prevalence of diabetes mellitus in 2019 is estimated to be 9.3% (463 million people).1 Diabetic retinopathy (DR) is microangiopathy characterized by capillary non- perfusion, microaneurysms (MAs), and retinal ischemia. 2It may cause many complications, such as diabetic macular edema (DME) and diabetic macular ischemia (DMI).3 Capillary ischemia decreases the nutrition of the retina and causes hypoxia which results in increased level of vascular endothelial growth factor (VEGF), which promotes angiogenic responses causing both neovascularization (proliferative diabetic retinopathy, PDR) and vascular permeability (macular edema).

Panretinal photocoagulation (PRP) by argon or diode laser is the standard treatment for proliferative diabetic retinopathy. It improves oxygenation to the ischemic retina. Destruction of the highly active photoreceptor cells is the suggested mechanism of action for PRP. Subsequently, production of vascular endothelial growth factor (VEGF), the key player in neovascularization process, is reduced leading to regression of new vessels.5

PDR eyes have an overall lower blood flow than normal or non-PDR eyes, parallel to the higher level of retinal ischemia and disease severity. With regression of these neovascular and shunt vessels following PRP, normalization of flow in the macula may reverse the ischemia and decrease the stimulus for new blood vessel formation. Closure of intraretinal microvascular abnormalities and neovascularization would theoretically increase overall resistance to flow and, combined with the constriction of the large vessel in response to increased oxygen in the inner retina, collectively decrease the overall blood flow.6 While most previous studies have explored the large vessel effects of PRP, the development of ocular coherence tomography angiography (OCTA) allowed the study of microvascular retinal changes in a detailed manner. It is a non-invasive modality that allows vascular mapping with high speed and quality and promotes visualization of vascular system in different retinal and choroidal levels. Several investigations have demonstrated the competence of OCTA in the quantification of microvascular density, choroidal flow area, and foveal avascular zone (FAZ) area in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes with PDR
* treatment-naive PDR diabetic patients diagnosed clinically and by the presence of neovascularization on optic disc (NVDs) or elsewhere (NVEs) on fluorescein angiography.

Exclusion Criteria:

* Patients with significant media opacity decreasing image quality

  -. Eyes with significant macular edema
* patients with glaucoma, uveitis, previous intraocular surgery, and history of previous treatment for diabetic retinopathy including anti-VEGF and laser
* patients with low signal strength index (SSI; <50)
* presence of 1 or more blink artifacts
* poor fixation leading to motion artifacts.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Measurement of vessel density | 6 months
  Measurement of vessel density at superficial, deep, and outer retina at base line, after 1 month, and after 6 months.
Measurement of retinal thickness | 6 months
  central retinal thickness at base line, after 1 month, and after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shawkat, Prof Dr, Study Director — Minia University Hospital; Mohamed Farouk, Prof Dr, Study Director — Minia University Hospital; Mohamed Salah, Doctor, Principal Investigator — Minia University Hospital; Asmaa Anwar, Doctor, Study Director — Minia University Hospital
Locations (1):
- Minia University Hospital, Minya, Egypt

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Adhi M, Brewer E, Waheed NK, Duker JS. Analysis of morphological features and vascular layers of choroid in diabetic retinopathy using spectral-domain optical coherence tomography. JAMA Ophthalmol. 2013 Oct;131(10):1267-74. doi: 10.1001/jamaophthalmol.2013.4321. PMID 23907153
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Miwa Y, Murakami T, Suzuma K, Uji A, Yoshitake S, Fujimoto M, Yoshitake T, Tamura Y, Yoshimura N. Relationship between Functional and Structural Changes in Diabetic Vessels in Optical Coherence Tomography Angiography. Sci Rep. 2016 Jun 28;6:29064. doi: 10.1038/srep29064. PMID 27350562
- [Background] Savage HI, Hendrix JW, Peterson DC, Young H, Wilkinson CP. Differences in pulsatile ocular blood flow among three classifications of diabetic retinopathy. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4504-9. doi: 10.1167/iovs.04-0077. PMID 15557461
- [Background] Cuypers MH, Kasanardjo JS, Polak BC. Retinal blood flow changes in diabetic retinopathy measured with the Heidelberg scanning laser Doppler flowmeter. Graefes Arch Clin Exp Ophthalmol. 2000 Dec;238(12):935-41. doi: 10.1007/s004170000207. PMID 11196354
- [Background] Ghassemi F, Fadakar K, Bazvand F, Mirshahi R, Mohebbi M, Sabour S. The Quantitative Measurements of Vascular Density and Flow Areas of Macula Using Optical Coherence Tomography Angiography in Normal Volunteers. Ophthalmic Surg Lasers Imaging Retina. 2017 Jun 1;48(6):478-486. doi: 10.3928/23258160-20170601-06. PMID 28613354
- [Background] Lee R, Wong TY, Sabanayagam C. Epidemiology of diabetic retinopathy, diabetic macular edema and related vision loss. Eye Vis (Lond). 2015 Sep 30;2:17. doi: 10.1186/s40662-015-0026-2. eCollection 2015. PMID 26605370
- [Derived] Abdelhalim AS, Abdelkader MFSO, Mahmoud MSE, Mohamed Mohamed AA. Macular vessel density before and after panretinal photocoagulation in patients with proliferative diabetic retinopathy. Int J Retina Vitreous. 2022 Mar 14;8(1):21. doi: 10.1186/s40942-022-00369-1. PMID 35287760